CLINICAL TRIAL: NCT02053090
Title: Complementary and Alternative Medicine (CAM) for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Scott Mist, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23AT006392 (NIH)
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Group Acupuncture; Group Education with Stretching; Nociceptive Reflex Testing; Pain; Sleep; Fatigue
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Education with Stretching (Active Comparator): Group Education with Stretching will receive 10 small group educational classes at the Oregon Health & Science University (OHSU), based on the book "Fibromyalgia (Biographies of Disease)." Each chapter of Fibromyalgia covers different aspects of the disease and its treatment including global, economic, and risk statistics; a timeline of key events in the study of fibromyalgia; common symptoms and diagnostic indicators; natural history of fibromyalgia; pharmacologic and non-pharmacologic treatments; associated disorders and syndromes; and impact of fibromyalgia at home, in the workplace and in society at large. Participants will be informed that they should not start additional treatments until the end of the study and complementary and alternative treatments won't be covered until the last session. Participants will also receive a digital video disk (DVD) covering stretching appropriate for fibromyalgia patients and will be asked to incorporate the DVD over the next 10 weeks.
  Interventions: Behavioral: Group Education and Stretching
- Group Acupuncture (Experimental): 20 treatments in 10 weeks will include individualized acupuncture in a group setting, dietary and lifestyle recommendations each based on the Traditional Chinese Medicine diagnosis (zhang fu) at the time of the visit.
  Interventions: Procedure: Group Acupuncture

INTERVENTIONS:
Behavioral: Group Education and Stretching
  Arms: Group Education with Stretching
Procedure: Group Acupuncture
  Arms: Group Acupuncture

SUMMARY:
This study is an acceptability and feasibility study of two adjunctive interventions: group education with stretching; and group acupuncture. The study population will be women with primary fibromyalgia who have not previously used acupuncture in the last 3 months. Both interventions will be 10 weeks in length and will be conducted at the Oregon Health & Science University. The primary hypothesis is that both arms will be acceptable and feasible in the study population.

ELIGIBILITY:
Inclusion Criteria:

1. Having met American College of Rheumatology (1990) criteria for the diagnosis of fibromyalgia
2. Having a primary Traditional Chinese Medicine (TCM) diagnosis of either Liver Qi Stagnation, Qi and Blood Stagnation, or Qi and Blood Deficiency
3. Female gender
4. Reported average pain of 5 or higher over last week on a scale of 0 to 10 with ten indicating higher pain.
5. Willingness to limit the introduction or change of any medications or treatment modalities for control of fibromyalgia symptoms during the study
6. No TCM in last 3 months (including acupuncture, Chinese herbs or herbal tea pills, tuina (Chinese massage), shiatsu (Japanese massage), qigong and Oriental food therapy)
7. Ability to travel to the intervention and testing sites up to two times weekly
8. Being over 18 and under 75 years of age, and
9. Capability of giving informed consent.

Exclusion Criteria:

1. Presence of a known coagulation abnormality, thrombocytopenia, or bleeding diathesis that may preclude the safe use of acupuncture;
2. Individuals with celiac disease
3. A score greater than 29 on the Beck Depression Inventory
4. Presence of concurrent autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, that causes pain and could potentially confound the analysis;
5. Routine daily use of narcotic analgesics or history of substance abuse;
6. Concurrent participation in other therapeutic trials;
7. Pregnant and nursing mothers (verification of pregnancy status will be determined via a urine test);
8. Severe psychiatric illnesses (current schizophrenia, major depression with suicidal ideation, substance abuse within two years);
9. Are undergoing disability determination, or are involved in litigation related to fibromyalgia
10. Any impairment, activity or situation that in the judgment of the PI would prevent satisfactory completion of the study protocol
11. Cognitive behavioral therapy in the last 6 months.
12. Non-fluency in English

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Treatment Participation Rate | 10 weeks
  Rates of treatment attendance in both arms

SECONDARY OUTCOMES:
Drop out rate | 10 and 14 weeks
  Drop out rates in both arms at weeks 10 and 14
Completion of Evaluation Rates | Weeks 0, 5, 10 and 14
  Completion rates of questionnaires and examinations in both arms
Fibromyalgia Impact Questionnaire Revised | Weeks 0, 5, 10, and 14
  Comparing overall score of the Fibromyalgia Impact Questionnaire - Revised between the two arms over time.
Nociceptive Reflex Testing | Weeks 0, 5, 10 and 14
  Nociceptive Reflex will be tested at weeks 0, 5, 10 and 14. Changes in nociceptive reflex will be compared within individuals and between arms.
Sleep Quality and Daily Activity | Weeks 0, 5, 10, and 14
  Sleep quality and daily activity will be measured using Actiwatch. Changes will be explored within individuals and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Mist, PhD, MAcOM, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States